CLINICAL TRIAL: NCT04925869
Title: Prospective Study of Cerebrovascular Accidents (CVA) in 3 French Cities (Besançon, Cayenne and Tours)
Acronym: AVCBCT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Centre Hospitalier Régional Universitaire de Tours (Other Government); Centre Hospitalier Régional Universitaire, Besançon (Unknown)
Responsible Party: Sponsor
Other Study IDs: AVC BCT
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Cerebrovascular Accident; Thrombolysis
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The hospitals of Besançon: Adult patients with MRI-confirmed CVA admitted to the hospitals of Besançon
  Interventions: Other: Observational study
- the hospitals of Cayenne: Adult patients with MRI-confirmed CVA admitted to the hospitals of Cayenne.
  Interventions: Other: Observational study
- the hospitals of Tours: Adult patients with MRI-confirmed CVA admitted to the hospitals of Tours.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
The objective of this study is to specify the typology of CVA in French Guiana by prospectively comparing consecutive strokes observed at each of the three study sites (Cayenne, Tours, Besançon)

DETAILED DESCRIPTION:
CVA is a public health problem that is managed in a codified manner by the Neurovascular Units (NU). In Cayenne, in the absence of a NU, strokes are managed directly in the emergency room by 24-hour telemedicine provided by the neurovascular team at the Besançon University Hospital. The vascular neurologist can perform a clinical examination remotely in a dedicated examination room and has access to magnetic resonance imaging by image transfer. The Tours and Besançon university hospitals each have a regional reference NU. The coordinating investigator of the study is the head of the neurology department of the Tours University Hospital, currently on an extended mission in Cayenne. The initial emergency management of a person with stroke who is hospitalized is comparable between the three regions studied.

Epidemiological studies show disparities in stroke mortality and vascular risk factors between French regions. The stroke mortality rate in French Guiana in 2013 (72 per 100 000 population per year) was twice that of metropolitan France. The standardized prevalence rate of diabetes in French Guiana is 7.1% of the population compared with 4.4% in metropolitan France, and the prevalence of hypertension is twice as high among women in the French Guiana West Indies compared with metropolitan France. There are twice as many obese persons (BMI>30) in Guyanese women compared with metropolitan France.

We propose a prospective observational study based on the following hypothesis:

The average age of stroke occurrence, its type (ischemic or hemorrhagic), the vascular territories involved, the vascular risk factors, and the pre-hospital and intra-hospital management times will be superimposable between two metropolitan regions but different in French Guyana.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of Cerebral Vascular Accident confirmed on MRI

Exclusion Criteria:

* Age under 18 years
* Absence of MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult patients with MRI-confirmed CVA admitted to the hospitals of Besançon, Cayenne, and Tours.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Describe the types of CVA and assess their risk factors on clinical, radiological and biological evidence | 3 months
  Clinical assessment of stroke (NIHSS score) and systematic collection of vascular risk factors (diabetes, hypertension, dyslipidemia, emboligic heart disease) Suspected mechanism (TOAST). Modified Rankin score

SECONDARY OUTCOMES:
Compare the time required for treatment between Cayenne, Besançon and Tours in the event of an indication for thrombolysis | 3 months
  Time to access care and management. The following will be specified: the time between the onset of symptoms and admission, MRI, and thrombolysis, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand De Toffol, PHD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, Guiana, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided